CLINICAL TRIAL: NCT01342731
Title: Effectiveness and Safety of Tigecycline for Therapy of Infections Caused by Multi-Drug Resistant Acinetobacter Baumannii
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Visanu Thamlikitkul, Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEU 003-11
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Antibiotic Resistant Infection
Keywords: Tigecycline; A.baumannii; Drug safety
MeSH Terms: interventions — Tigecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tigecycline (Experimental): Tigecycline 100 mg of tigecycline intravenous infusion for 30 minutes followed by 50 mg every 12 hours for 7 to 14 d
  Interventions: Drug: Tigecycline

INTERVENTIONS:
Drug: Tigecycline — 100 mg of tigecycline intravenous infusion for 30 minutes followed by 50 mg every 12 hours for 7 to 14 days.
  Other Names: Tygacil

SUMMARY:
30 adult hospitalized patients who have infections due to MDR Acinetobacter baumannii will be enrolled. The eligible patients will receive 100 mg of tigecycline intravenous infusion for 30 minutes followed by 50 mg every 12 hours for 7 to 14 days. Clinical outcomes on effectiveness and safety will be evaluated on daily basis up to 28 days. Follow-up culture of clinical specimen from the site of infection will be obtained on day 3 and at the end of tigecycline therapy. Clinical response is classified as cure, improvement, failure, relapse, death. Microbiological outcome is assessed at the end of treatment and classified as eradication, persistence, colonization, and superinfection. Adverse events, overall 28-day mortality and infection-related mortality will be determined. Length of stay will also be determined.

DETAILED DESCRIPTION:
Objectives:

To determine effectiveness and safety of tigecycline for therapy of hospitalized patients with infections due to MDR A. baumannii.

Study Design Open label phase IV study

Sample Size:

It is estimated that a favorable response rate in patients infected with MDR A. baumannii who received tigecycline is 60% +/- 20% with 5% type I error. Therefore the estimated sample size is 24 patients. This study will enroll 30 patients in order to compensate for some patients who may not be available to have a complete follow up.

Study Procedures:

All eligible patients will be identified through the pharmacy database and microbiology database on daily basis. The investigator will obtain written consent from each potential patient. Consent must be documented by the patient's dated signature on a consent form along with the dated signature of the person conducting the consent discussion. If the patient is in the state that can not make decision, the written consent of a parent, legal guardian or legal representative must be obtained. Intervention: The eligible patients will receive 100 mg of tigecycline intravenous infusion for 30 minutes followed by 50 mg every 12 hours for 7 to 14 days.

Evaluation/Follow - Up:

Clinical outcomes on effectiveness and safety will be evaluated on daily basis up to 28 days. Follow-up culture of clinical specimen from the site of infection will be obtained on day 3 and at the end of tigecycline therapy. Clinical response is classified as cure, improvement, failure, relapse, death. Microbiological outcome is assessed at the end of treatment and classified as eradication, persistence, colonization, and superinfection. Adverse events, overall 28-day mortality and infection-related mortality will be determined. Length of stay will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male or female aged 18 years or older
* Has documented infection due to A. baumannii resistant to cephalosporins, beta-lactams/ beta-lactamase inhibitors, aminoglycosides, fluoroquinolones and carbapenems
* Willing to join the study by signing a written informed consent form

Exclusion Criteria:

* Pregnant or lactating woman
* Has contraindication for receiving tigecycline such as allergy to tetracycline
* Has received colistin for more than 24 hours
* Unable to receive tigecycline monotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | at the end of therapy (up to 28 days)
  Clinical response is classified as cure, improvement, failure, relapse, death.

SECONDARY OUTCOMES:
Microbiological outcomes | At the end of therapy (up to 28 days)
  Microbiological outcome is classified as eradication, persistence, colonization, and superinfection.

CONTACTS AND LOCATIONS:
Overall Officials: Visanu Thamlikitkul, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand